CLINICAL TRIAL: NCT02462395
Title: Anodal Transcranial Direct Stimulation (tDCS) of the Anterior Cingulate Gyrus for the Treatment of Chronic Cluster Headache: a Pilot Trial.
Brief Title: Anodal Transcranial Direct Stimulation (tDCS) for the Treatment of Chronic Cluster Headache
Acronym: ANODECCH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean Schoenen, Honorary Full Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANODECCH
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cefaly tDCS (Experimental): Sponge-electrodes (5 x 7 cm) will be postioned at Fz (anode) and over the spinous process of C7 (cathode). Stimulation intensity will be set to 2 mA.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Sponge-electrodes (5 x 7 cm) will be postioned at Fz (anode) and over the spinous process of C7 (cathode). Stimulation intensity will be set to 2 mA.
  A first group of CCH patients will have to apply the neurostimulation outside of an attack every day for 20 minutes during 4 weeks. A second group will use the tDCS device everyday for 8 weeks.
  Adherence to the treatment will be evaluated by monitoring the time during which the device is switched on via an in-built software.
  Other Names: tDCS Cefaly Technology°.

SUMMARY:
Cluster headache is a primary headache that chiefly affects young men, and is less common than migraine. This disease can have devastating consequences due to the pain intensity (it is also called "suicide headache"), to the side effects of the drug preventive therapies, and to the resistance of some subtypes of the headache to all existing medications.

Recent studies suggest that cluster headache could be associated with a decrease of the activity of frontal areas involved in descending pain control, in particular the subgenual anterior cingulate cortex. The aim of this pilot study is to activate these areas with a non-invasive neurostimulation technique, called transcranial direct current stimulation, as a preventive treatment for cluster headache sufferers.

DETAILED DESCRIPTION:
Cluster headache affects 0.1%-0.25% of the general population, but its prevalence may be underestimated. It is a primary headache disorder with a higher prevalence in young males, characterized by attacks of severe unilateral periorbital/temporal pain with autonomic symptoms (ie lacrimation, nasal congestion, eyelid edema, Horner's…) and agitation, lasting 15 to 180 minutes and occurring periodically in bouts (clusters) in about 90% of patients (episodic cluster headache or ECH, ICHD-III criteria 3.1.1).In 10% of patients there is no sustained spontaneous remission for long periods, which defines chronic cluster headache (CCH, ICHD-III criteria 3.1.2).

The pathophysiology of cluster headache is not completely understood, but neuroimaging studies clearly suggest that activation of the ipsilateral postero-ventral hypothalamus plays a seminal role during the attack. Recent findings suggest that prefrontal areas may be dysfunctioning in cluster headache patients. The investigator shave shown in CCH patients that the beneficial effects of ONS are associated with activation of the subgenual anterior cingulate cortex, an area responsible for descending pain-control. Transcranial direct current stimulation (tDCS) allows activating the underlying cortex and connected subcortical structures under the anode or inhibiting them under the cathode. tDCS was used as a therapeutic strategy in various neurological disorders, chronic pain disorders and depression. Because of its non-invasiveness, It is of particular interest in primary headaches where various brain areas are known to function abnormally even between headache attacks. It has been tested in migraine but not in cluster headache.

In a recent study, the investigators have shown that anodal tDCS over the visual cortex is able to modify visual evoked potentials in healthy volunteers and migraineurs, and after a 2-month treatment of 2 weekly sessions to significantly decrease attack frequency in episodic migraine.

CCH patients will have to apply the neurostimulation outside of an attack every day for 20 minutes during 4 to 8 weeks.

Adherence to the treatment will be evaluated by monitoring the time during which the device is switched on via an in-built software.

ELIGIBILITY:
Inclusion Criteria:

* Main inclusion criteria for CCH: preventive CH therapy stable for a least 2 months, retrospective 4-week headache baseline diary showing at least 4 attacks/week on average

Exclusion Criteria:

* No other significant medical or psychiatric disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Reduction of weekly cluster headache attack frequency during and following tDCS treatment in CCH patients. | 4 to 8 weeks
  Analysis of the headache diary

SECONDARY OUTCOMES:
reduction of intensity of CH attacks | 4 to 8 weeks
  Analysis of the headache diary
reduction of duration of CH attacks | 4 to 8 weeks
  Analysis of the headache diary
reduction of acute medication intake | 4 to 8 weeks
  Analysis of the headache diary
modification of the nociceptive blink reflex | 4 to 8 weeks
modification of pain thresholds | 4 to 8 weeks
  using quantitative sensory testing

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Magis, MD, Principal Investigator — University of Liege
Locations (1):
- CHR Citadelle, Liège, Liege, Belgium